CLINICAL TRIAL: NCT06073366
Title: Long-term Surveillance of Patients With Venous Thromboembolism: a Nationwide Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lu Hua, Chief Physician, China National Center for Cardiovascular Diseases
Other Study IDs: 2022-I2M-C&T-B-040
Record Dates: First submitted 2023-07-17; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to establish a prospective nationwide cohort of venous thromboembolism. The main questions it mains to answer are:

* Which patients with venous thromboembolism should accept long-term anticoagulation therapy?
* Mechanism and prognosis of venous thromboembolism. Participants will receive yearly follow-ups through telephone, hospitalization, or outpatient care.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE), including deep venous thrombosis and pulmonary embolism, is a class of diseases with strong occultation, high mortality, and a high recurrence rate.Long-term anticoagulant therapy can reduce the risk of recurrence. Although long-term anticoagulation can reduce the risk of VTE recurrence, it will also increase the risk of major bleeding and the economic burden of long-term anticoagulation. Therefore, stratifying the risk of VTE recurrence and preventing recurrence with accurate anticoagulant therapy is an urgent problem in VTE management.

Investigators will establish a prospective nationwide cohort of VTE, develop a unified follow-up plan, and conduct whole-life follow-up management for patients. Demographic, clinical, imaging, laboratory indicators, gene, and other information of patients will be collected. A VTE patient database with complete clinical phenotype data, genetic data, and biological samples will be established.

Investigators will construct a VTE recurrence risk prediction model based on Chinese data to provide clinical decision suggestions for clinicians to select appropriate individualized anticoagulant duration according to risk stratification. VTE patients with low recurrence risk could avoid long-term anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18.
* Patients diagnosed with venous thromboembolism.

Exclusion Criteria:

* Pregnant or lactating women
* Patients with active tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients diagnosed with venous thromboembolism will be eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence | through study completion, an average of 1 year
  recurrence of venous thromboembolism

SECONDARY OUTCOMES:
Bleeding episode | through study completion, an average of 1 year
  The definition of bleeding episode is consistent with the guideline of international society thrombosis & hemostasis
All-cause death | through study completion, an average of 1 year
  All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hua, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khan F, Rahman A, Carrier M, Kearon C, Weitz JI, Schulman S, Couturaud F, Eichinger S, Kyrle PA, Becattini C, Agnelli G, Brighton TA, Lensing AWA, Prins MH, Sabri E, Hutton B, Pinede L, Cushman M, Palareti G, Wells GA, Prandoni P, Buller HR, Rodger MA; MARVELOUS Collaborators. Long term risk of symptomatic recurrent venous thromboembolism after discontinuation of anticoagulant treatment for first unprovoked venous thromboembolism event: systematic review and meta-analysis. BMJ. 2019 Jul 24;366:l4363. doi: 10.1136/bmj.l4363. PMID 31340984
- [Background] Rodger MA, Kahn SR, Wells PS, Anderson DA, Chagnon I, Le Gal G, Solymoss S, Crowther M, Perrier A, White R, Vickars L, Ramsay T, Betancourt MT, Kovacs MJ. Identifying unprovoked thromboembolism patients at low risk for recurrence who can discontinue anticoagulant therapy. CMAJ. 2008 Aug 26;179(5):417-26. doi: 10.1503/cmaj.080493. PMID 18725614
- [Background] Eichinger S, Heinze G, Jandeck LM, Kyrle PA. Risk assessment of recurrence in patients with unprovoked deep vein thrombosis or pulmonary embolism: the Vienna prediction model. Circulation. 2010 Apr 13;121(14):1630-6. doi: 10.1161/CIRCULATIONAHA.109.925214. Epub 2010 Mar 29. PMID 20351233
- [Background] Tosetto A, Iorio A, Marcucci M, Baglin T, Cushman M, Eichinger S, Palareti G, Poli D, Tait RC, Douketis J. Predicting disease recurrence in patients with previous unprovoked venous thromboembolism: a proposed prediction score (DASH). J Thromb Haemost. 2012 Jun;10(6):1019-25. doi: 10.1111/j.1538-7836.2012.04735.x. PMID 22489957
- [Background] Franco Moreno AI, Garcia Navarro MJ, Ortiz Sanchez J, Martin Diaz RM, Madronal Cerezo E, de Ancos Aracil CL, Cabello Clotet N, Perales Fraile I, Gimeno Garcia S, Montero Hernandez C, Zapatero Gaviria A, Ruiz Giardin JM. A risk score for prediction of recurrence in patients with unprovoked venous thromboembolism (DAMOVES). Eur J Intern Med. 2016 Apr;29:59-64. doi: 10.1016/j.ejim.2015.12.010. Epub 2016 Jan 8. PMID 26775136
- [Background] Le Gal G, Kovacs MJ, Bertoletti L, Couturaud F, Dennie C, Hirsch AM, Huisman MV, Klok FA, Kraaijpoel N, Mallick R, Pecarskie A, Pena E, Phillips P, Pichon I, Ramsay T, Righini M, Rodger MA, Roy PM, Sanchez O, Schmidt J, Schulman S, Shivakumar S, Trinh-Duc A, Verdet R, Vinsonneau U, Wells P, Wu C, Yeo E, Carrier M; SSPE Investigators. Risk for Recurrent Venous Thromboembolism in Patients With Subsegmental Pulmonary Embolism Managed Without Anticoagulation : A Multicenter Prospective Cohort Study. Ann Intern Med. 2022 Jan;175(1):29-35. doi: 10.7326/M21-2981. Epub 2021 Nov 23. PMID 34807722